CLINICAL TRIAL: NCT02221583
Title: A Multicenter Pilot Study to Determine the Pharmacokinetics of Astagraf XL, Prograf and Mycophenolate Mofetil in Renal Transplant Candidates Who Have Undergone Laparoscopic Sleeve Gastrectomy
Brief Title: Pharmacokinetics of Immunosuppressants in Renal Transplant Candidates Who Have Undergone Laparoscopic Sleeve Gastrectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Principal Investigator, Tayyab Diwan, Assistant Professor of Surgery, University of Cincinnati
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: ASTA-14B02
Record Dates: First submitted 2014-08-13; First posted 2014-08-20 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: End Stage Renal Disease
Keywords: End stage renal disease; Renal transplant candidate; Laparoscopic sleeve gastrectomy; Immunosuppressants
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Astagraf XL + Mycophenolate mofetil then cross over to Prograf + Mycophenolate
  Interventions: Drug: Astagraf XL; Drug: Prograf; Drug: Mycophenolate mofetil
- Group 2 (Experimental): Prograf + Mycophenolate mofetil then cross over to Astagraf XL + Mycophenolate
  Interventions: Drug: Astagraf XL; Drug: Prograf; Drug: Mycophenolate mofetil

INTERVENTIONS:
Drug: Astagraf XL — Two PK profiles will be obtained in each subject. Each subject will receive either Astagraf XL 8mg daily or Prograf® 4mg every 12 hours in combination with MMF 1000mg every 12 hours. A full 24 hour PK profile will be constructed. After at least a one week washout period, the patient will be crossed over to the alternative tacrolimus formulation (Astagraf XL or Prograf®) in combination with MMF 1000mg every 12 hours and the PK profile repeated.
  Other Names: Tacrolimus sustained release
Drug: Prograf — Two PK profiles will be obtained in each subject. Each subject will receive either Astagraf XL 8mg daily or Prograf® 4mg every 12 hours in combination with MMF 1000mg every 12 hours. A full 24 hour PK profile will be constructed. After at least a one week washout period, the patient will be crossed over to the alternative tacrolimus formulation (Astagraf XL or Prograf®) in combination with MMF 1000mg every 12 hours and the PK profile repeated.
  Other Names: Tacrolimus
Drug: Mycophenolate mofetil — Two PK profiles will be obtained in each subject. Each subject will receive either Astagraf XL 8mg daily or Prograf® 4mg every 12 hours in combination with MMF 1000mg every 12 hours. A full 24 hour PK profile will be constructed. After at least a one week washout period, the patient will be crossed over to the alternative tacrolimus formulation (Astagraf XL or Prograf®) in combination with MMF 1000mg every 12 hours and the PK profile repeated.
  Other Names: Cellcept

SUMMARY:
The purpose of this study is to evaluate how quickly and to what extent different immunosuppressants are absorbed into the blood (this is called pharmacokinetics) in renal transplant candidates who have undergone a laparoscopic sleeve gastrectomy. The immune system is the body's defense against diseases. It also attacks "foreign" tissues such as a transplanted kidney. Immunosuppressant medications such as Astagraf sustained release (XL), Prograf, and mycophenolate mofetil may be given to suppress the immune system following kidney transplantation and prevent rejection of a transplanted kidney. This study is being performed to determine if patients who undergo laparoscopic sleeve gastrectomy need different doses of immunosuppressant medications.

DETAILED DESCRIPTION:
Investigators propose a single dose, cross over pharmacokinetic study of Astagraf XL and Prograf® in combination with MMF in RTx candidates that have undergone LSG. Subjects at least three months post LSG and pre-renal transplant will undergo preliminary screening. The study population will consist of 24 male and female subjects, ≥ 18 years old from UC Health University Hospital and The Christ Hospital who meet the inclusion/exclusion criteria.

Two PK profiles will be obtained in each subject. Each subject will receive either Astagraf XL 8mg daily or Prograf® 4mg every 12 hours in combination with MMF 1000mg every 12 hours. A full 24 hour PK profile will be constructed. After at least a one week washout period, the patient will be crossed over to the alternative tacrolimus formulation (Astagraf XL or Prograf®) in combination with MMF 1000mg every 12 hours and the PK profile repeated. The immunosuppressants chosen reflect the regimen most commonly prescribed to transplant recipients.

Subjects participating in the study will have pharmacokinetic blood samples drawn over a 24 hour time period in order to determine the AUC, Tmax, Cmax, and half-life of tacrolimus, MMF and their metabolites. Samples would be drawn prior to dosing (C0) and at 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 12.5, 13, 14, 15, 16, 18, 20 and 24 hours post dosing (18 time points) by venipuncture or IV.

This study proposal represents a simple and expeditious method to achieve PK information in patients that have undergone LSG. If desired, study could be expanded to evaluate PK in additional patient groups such as pre and post LSG and/or pre and post renal transplant. The exact sample collection time will be recorded in the case report form. All deviations from the scheduled sampling time of more than 5 minutes for the first 4 hours after the AM dose (predose-4 hr) and first 4 hours of the PM dose (12 hr-16 hr), and more than 10 minutes for all remaining samples (6 hr-8 hr; 18 hr-24 hr) will be reported as a protocol deviation.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male patient aged > 18 years old.
2. ESRD patient (on dialysis or preemptive) who is a potential candidate for kidney transplantation
3. Undergone laparoscopic sleeve gastrectomy procedure > 3 months prior to enrollment.
4. Subjects have signed and dated the informed consent to participate in the study.

Exclusion Criteria:

1. Patients taking a drug known to interact with Astagraf XL, Prograf®, or MMF.
2. Patients that have an allergy to Astagraf XL, Prograf®, or MMF.
3. Patients currently taking Astagraf XL, Prograf®, or MMF.
4. Post-surgical leak complication
5. Patients failing to adhere to post laparoscopic sleeve gastrectomy follow-up recommendations and clinic visits
6. Patients with any severe medical condition requiring acute or chronic treatment that in the investigator's opinion would interfere with study participation.
7. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive laboratory test
8. Currently taking or planning to initiate of any medications that could interfere with tacrolimus and/or mycophenolate blood levels, including over the counter (OTC) medications, herbal supplements, grapefruit or grapefruit juice.
9. Subjects who have been exposed to an investigational therapy within 30 days prior to enrollment or 5 half-lives of the investigational product, whichever is greater.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-05; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Area Under Curve (AUC) | Prior to dosing (CO), and at 1, 1.5, 2, 2.5, 3, 4, 6, 8,12, 12.5, 13, 14, 15, 16, 18, 20 and 24 hours post dosing
  AUC of tacrolimus, MMF and their metabolites will be measured at 18 timepoints within 24 hour period on Study Day 1 and Day 8
Maximum concentration (Cmax) | Prior to dosing (CO), and at 1, 1.5, 2, 2.5, 3, 4, 6, 8,12, 12.5, 13, 14, 15, 16, 18, 20 and 24 hours post dosing
  Cmax of tacrolimus, MMF and their metabolites will be measured at 18 timepoints within 24 hour period on Study Day 1 and Day 8
Time to maximum concentration (Tmax) | Prior to dosing (CO), and at 1, 1.5, 2, 2.5, 3, 4, 6, 8,12, 12.5, 13, 14, 15, 16, 18, 20 and 24 hours post dosing
  Tmax of tacrolimus, MMF and their metabolites will be measured at 18 timepoints within 24 hour period on Study Day 1 and Day 8
Half life (T 1/2) | 24 hours
  Half-life of tacrolimus, MMF and their metabolites will be measured at 18 timepoints within 24 hour period on Study Day 1 and Day 8

SECONDARY OUTCOMES:
Adverse events (serious and non-serious) | Study Day 1 and Day 8
  All serious adverse events and non-serious adverse events as reported by the subject will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Tayyab Diwan, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Diwan TS, Lichvar AB, Leino AD, Vinks AA, Christians U, Shields AR, Cardi MA, Fukuda T, Mizuno T, Kaiser T, Woodle ES, Alloway RR. Pharmacokinetic and pharmacogenetic analysis of immunosuppressive agents after laparoscopic sleeve gastrectomy. Clin Transplant. 2017 Jun;31(6). doi: 10.1111/ctr.12975. Epub 2017 May 2. PMID 28342282